CLINICAL TRIAL: NCT06552936
Title: Combination Therapy Effect of Laser on Wound Healing and Bone Regeneration of Dental Sockets
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sharif Medical Research Center (Other)
Collaborators: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Amna Nauman, Professor, Sharif Medical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SMDC/SMRC/242-22
Record Dates: First submitted 2024-08-09; First posted 2024-08-14 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Tooth Extraction
Keywords: Tooth socket, Laser, wound healing, bone regeneration, pain
MeSH Terms: conditions — Pain | interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Low level laser therapy (LLLT) (Experimental): The LLLT phase will be done with an uninitiated 300-micron tip at 0.5 W in a CW. For this phase, the tip will be kept apart from the targeted tissue by 1mm in the scanning motion.
  Interventions: Other: Diode Laser 980 nm.
- High intensity laser therapy (HILT) (Experimental): HILT will be done directly after extraction when the extraction socket is filled with blood (without oozing). It will be conducted with the help of an un-initiated 300-micron tip running at the 2-watt (W) power output. It will be in a continuous emission mode (CW).
  Interventions: Other: Diode Laser 980 nm.
- Low level laser therapy+ high intensity laser therapy (Experimental): The patient will receive a combination of LLLT and HILT.
  Interventions: Other: Diode Laser 980 nm.
- Control (Sham Comparator): The patient will have the identical treatment as the experimental group but with the laser device in the non-activated phase.
  Interventions: Other: Diode Laser 980 nm.

INTERVENTIONS:
Other: Diode Laser 980 nm. — A Diode laser is commonly used in simple surgical procedures on soft tissue, such as skin or mucosa. Its tip can work when non-activated, causing inductive effects, and when activated, it causes the ablation of soft tissue.

SUMMARY:
The goal of this clinical trial is to learn if the laser works to improve wound healing and bone regeneration after tooth extraction. The main question it aims to answer is:

Does laser therapy improve wound healing and bone regeneration after tooth extraction?

Researchers will compare a laser to sham laser therapy to see if the laser enhances wound healing and bone regeneration.

Participants will:

Have exposure to laser or sham laser therapy immediately after tooth extraction Record their pain intensity on days 2, 4, 6 and 14 Visit the clinic after 10 days for follow-up Again, visit the clinic after 4 months for evaluation

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years old, regardless of gender
* Non-traumatic tooth extraction of the lower jaw is indicated
* Willing for dental implant surgery
* Dental appointments are available at the study place
* Absence of active infection at the extraction site
* Signed informed permission is provided.

Exclusion Criteria:

* Pregnant, lactating, and menopausal women
* Smokers
* Those having head and neck radiotherapy
* Those with any sort of acute infection (e.g., periodontal abscess), immune deficiency, or metabolic conditions such as diabetes mellitus and osteoporosis
* Patients will also be eliminated if they have a complication during surgery, such as bleeding or operational difficulties, or if the procedure takes longer than 90 minutes.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Wound healing will be assessed in both the experimental and control groups. | 1 year
  Wound healing will be assessed using the Landry, Turnbull, and Howley index after 7 days, and a score will be given ranging from 1 to 5, where 1 indicates very poor healing, and 5 indicates excellent healing. (score range: 1-very poor, 2-poor, 3-good, 4-very good, 5-excellent)
Bone regeneration will be assessed in both the experimental and control groups. | 1 year
  A postoperative cone beam computed tomography (CBCT) will be taken immediately after extraction, followed by a CBCT 4 months after extraction. The immediate CBCT will be done to study the density of healthy bone in the apical region of the extracted tooth socket. This value will serve as the baseline for further assessment. The density obtained will then be compared with the bone formed at the end of 4 months in the extraction socket with and without laser therapy. Taking mean readings in the grayscale measurements from the periapical region will allow for the calculation of bone density.

SECONDARY OUTCOMES:
Pain intensity will be measured in both the experimental and control groups. | 1 year
  The Visual Analogue Scale (VAS) will assess pain intensity at post-extraction days 2, 4, 6, and 14. It consists of a 10 cm line with two endpoints representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). VAS is a system that classifies a score of 1 to 4 (on a 0-10 scale) as mild pain, 5 to 6 as moderate pain, and 7 to 10 as severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Amna N Khan, MPhil, Principal Investigator — Sharif Medical and Dental College
Locations (2):
- Pakistan (2):
  - Sharif Medical and Dental College, Lahore, Punjab Province
  - Sharif Medical and Dental College, Lahore

IPD SHARING:
Plan to Share IPD: No